CLINICAL TRIAL: NCT07330713
Title: Platelet-Rich Plasma for Acute Nonarteritic Anterior Ischemic Optic Neuropathy: A Prospective Randomized Controlled Study
Acronym: PRP-NAION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Gamze Uçan Gündüz, Associate Professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-21/36
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Nonarteritic Anterior Ischemic Optic Neuropathy
Keywords: nonarteritic anterior ischemic optic neuropathy, platelet-rich plasma, subtenon injection
MeSH Terms: conditions — Optic Neuropathy, Ischemic

STUDY DESIGN:
Intervention Model Description: Eligible participants are randomly assigned to one of two parallel groups. One group receives posterior subtenon autologous platelet-rich plasma injections, while the control group is managed with observation alone. Participants remain in their assigned groups throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Treatment Group (Experimental): Participants receive posterior subtenon autologous platelet-rich plasma injections in addition to standard clinical follow-up.
  Interventions: Biological: Autologous Platelet-Rich Plasma (PRP)
- Control Group (No Intervention): Participants are managed with observation alone and receive no interventional treatment.

INTERVENTIONS:
Biological: Autologous Platelet-Rich Plasma (PRP) — Autologous platelet-rich plasma is prepared from the participant's own blood and administered via posterior subtenon injection at scheduled visits.
  Arms: PRP Treatment Group

SUMMARY:
This prospective randomized clinical study aims to evaluate the efficacy and safety of autologous platelet-rich plasma (PRP) injection in patients with acute non-arteritic anterior ischemic optic neuropathy (NAION). Eligible patients are randomly assigned to receive posterior subtenon PRP injections or to an observation-only control group. The PRP group receives injections at baseline and during follow-up. Comprehensive ophthalmologic evaluations, including best-corrected visual acuity, visual field testing, and retinal nerve fiber layer thickness measurements, are performed at baseline and scheduled follow-up visits. The primary outcomes include changes in visual function and structural optic nerve parameters, as well as the incidence of treatment-related adverse events.

DETAILED DESCRIPTION:
This prospective randomized clinical study is designed to evaluate the efficacy and safety of posterior subtenon autologous platelet-rich plasma (PRP) injection in patients diagnosed with acute non-arteritic anterior ischemic optic neuropathy (NAION). Patients meeting the inclusion criteria are enrolled and randomly assigned, using computer-assisted randomization, to either the PRP treatment group or an observation-only control group.

Patients in the PRP group receive posterior subtenon injections of autologous PRP at baseline and during scheduled follow-up visits. The control group is managed with observation alone and receives no interventional treatment. All participants undergo comprehensive ophthalmologic examinations at baseline and at predefined follow-up visits, including assessments of best-corrected visual acuity, visual field testing, and retinal nerve fiber layer thickness measurements obtained by optical coherence tomography.

Patients are followed longitudinally to assess changes in functional and structural optic nerve parameters, as well as to monitor for any ocular or systemic adverse events related to the intervention. Safety evaluations are performed at each follow-up visit throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute non-arteritic anterior ischemic optic neuropathy (NAION) based on clinical history and ophthalmologic examination

Acute, painless vision loss and/or visual field defect

Symptom onset within 14 days prior to enrollment

Age 40 years or older

Ability to cooperate with best-corrected visual acuity and visual field examinations

Willingness and ability to complete all follow-up visits (weeks 1, 3, 6, 8, and 16)

Provision of written informed consent

Exclusion Criteria:

* Arteritic anterior ischemic optic neuropathy

Posterior ischemic optic neuropathy

Age under 40 years

Presence of concomitant ocular diseases that could affect visual outcomes (e.g., glaucoma, diabetic macular edema, retinal dystrophy)

Presence of neurological diseases that may affect the optic nerve (e.g., demyelinating disease, intracranial or intraorbital mass)

Inability to cooperate with visual acuity or visual field testing

Presence of systemic hematological disorders that could interfere with platelet-rich plasma preparation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) | Baseline (Week 0) to Week 16
  Change in best-corrected visual acuity from baseline (week 0) to week 16, measured in logarithm of the minimum angle of resolution (logMAR) units using standard visual acuity charts.

SECONDARY OUTCOMES:
Change in Visual Field Mean Deviation (MD) and Visual Field Index (VFI) | Baseline (Week 0) to Week 16
  Change in visual field mean deviation (MD) and visual field index (VFI) measured by automated perimetry (Humphrey Field Analyzer 30-2) from baseline to week 16.
Change in Peripapillary Retinal Nerve Fiber Layer (RNFL) Thickness | Baseline (Week 0) to Week 16
  Change in global and sectoral peripapillary retinal nerve fiber layer thickness measured by spectral-domain optical coherence tomography (OCT) from baseline to week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ucan Gündüz, MD, Principal Investigator — Uludag University, Department of Ophthalmology; Selim Doganay, MD, Principal Investigator — Uludag University, Department of Ophthalmology
Locations (1):
- Uludag University, Department of Ophthalmology, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No